CLINICAL TRIAL: NCT05445076
Title: An International, Multicenter, Double-Blind, Randomized Placebo-Controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of BCD-180 in Patients With Axial Spondyloarthritis
Brief Title: Study of the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of BCD-180 in Patients With Axial Spondyloarthritis
Acronym: ELEFTA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-180-2
Record Dates: First submitted 2022-06-03; First posted 2022-07-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-06

CONDITIONS: Axial Spondyloarthritis
Keywords: biologics; axial spondyloarthritis; monoclonal antibodies; TRBV9
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCD-180, low dose (Experimental): Subjects in this arm will receive BCD-180 low dose infusions
  Interventions: Biological: anti-TRBV9 monoclonal antibody, low dose
- BCD-180, high dose (Experimental): Subjects in this arm will receive BCD-180 high dose infusions
  Interventions: Biological: anti-TRBV9 monoclonal antibody, high dose
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo till the assessment of the primary endpoint and then will be switched to BCD-180 low dose
  Interventions: Biological: anti-TRBV9 monoclonal antibody, low dose; Other: placebo

INTERVENTIONS:
Biological: anti-TRBV9 monoclonal antibody, low dose — infusion
  Arms: BCD-180, low dose; Placebo
Biological: anti-TRBV9 monoclonal antibody, high dose — infusion
  Arms: BCD-180, high dose
Other: placebo — infusion
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy, safety, immunogenicity, pharmacokinetics and pharmacodynamics of two doses of study drug (BCD-180) in comparison with placebo in patients with active radiographic axial spondyloarthritis (axSpA). The study will include HLA-B27+ patients with radiographic axSpA who had no response to prior therapy with Non-steroidal anti-inflammatory drugs (NSAIDs), have not received biologic therapy or targeted Disease-modifying antirheumatic drugs (DMARDs).

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria will be randomized in 3 groups to receive one of two studied doses of BCD-180 or placebo.

After the primary endpoint assessment subjects in placebo group will be switched to BCD-180 in minimal studied dose. After the completion of the main period of the study in each of the BCD-180 groups subjects who meet the criterion of non-active radiographic axSpA (ASDAS-CRP <1.3 at two subsequent visits) will be subjected to repeated randomization in two groups for the use of two different dosing regimens. Subjects of the Placebo group will continue to receive BCD-180 infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form for participation in the study.
2. Men and women aged 18 to 65 years inclusive at the time of signing the Informed Consent Form.
3. An established diagnosis of ankylosing spondylitis according to the modified New York classification criteria (van der Linden et al. 1984).
4. Sacroiliitis (bilateral ≥ grade 2 or unilateral grade 3-4) based on central review of radiographs.
5. Positive ASAS criteria for axial spondyloarthritis (Rudwaleit et al. 2009).
6. Duration of back pain ≥3 months and age of onset of back pain <45 years.
7. Positive HLA-B27 test.
8. Active disease at screening and at the Randomization Visit, based on both of the following criteria:

   * BASDAI ≥4,
   * back pain NRS score ≥4 (BASDAI question 2).
9. CRP level ≥5 mg/mL at screening.
10. At least one of the following criteria, as assessed by the investigator:

    1. Inadequate response to NSAID therapy defined as an insufficient response to NSAID therapy at a therapeutic dose for at least 4 weeks, or an insufficient response to therapy with two NSAIDs at the maximum allowed dose with a total duration of therapy of at least 4 weeks;
    2. Contraindications for NSAID therapy;
    3. Intolerance to more than one NSAID.
11. For subjects continuing to receive NSAIDs or COX-2 inhibitors: the dose of the drug should be stable for at least 14 days prior to Visit 1/Week 0.
12. For women: a negative pregnancy test at screening (the test is not performed in women who have been postmenopausal for at least 2 years or are surgically sterile) .
13. The ability of the subject, in the opinion of the investigator, to follow the protocol procedures.
14. Willingness of subjects and their sexual partners of childbearing potential to use reliable methods of contraception from the date of signing the ICF, throughout the study, and for 8 weeks after the last administration of the test drug/placebo. This requirement does not apply to subjects who have had operative sterilization and women who have been postmenopausal for more than 2 years. Reliable methods of contraception include the use of one barrier method in combination with one of the following in the female partner: spermicides, intrauterine device, oral contraceptives.
15. For subjects of childbearing potential (from the ICF signing, throughout the study, and for 8 weeks after the last infusion of the test drug/placebo):

    * no egg donation for female subjects;
    * no sperm donation for male subjects.

Exclusion Criteria:

1. Total ankylosis of the spine defined by the presence of syndesmophytes in ≥3 adjacent vertebral segments based on central review of radiographs.
2. Age less than 18 years at disease onset.
3. Refusal to take NSAIDs for the treatment of AS for any subjective reasons that do not have a clinical justification.
4. Use of the following medicines/procedures:

   * at any time before signing the ICF: use of any monoclonal antibodies or their fragments for any indication;
   * at any time before signing the ICF: total irradiation of the lymphatic system;
   * at any time before signing the ICF: bone marrow transplantation, including transplantation of stem and hematopoietic cells for any indication;
   * at any time before signing the ICF: splenectomy;
   * within 8 weeks before signing the ICF: treatment with immunoglobulins;
   * within 12 months before signing the ICF: use of immunosuppressants. Exception: glucocorticoids. A subject receiving glucocorticoids may be included in the study provided that the daily dose of glucocorticoids is ≤10 mg/day (calculated with reference to prednisolone) and was stable for at least 4 weeks prior to the Randomization Visit.
   * within 4 weeks before signing the ICF and during the screening period: use of synthetic DMARDs and thiopurines, including, but not limited to: 6-mercaptopurine, azathioprine, and others.

   Exception: the medicinal products listed below if their dose was stable for 4 weeks before signing the ICF and during the screening period:
   * methotrexate orally or parenterally at a dose not exceeding 25 mg/week, provided that therapy was started at least 8 weeks before signing the ICF;
   * 5-aminosalicylic acid and its derivatives, including sulfasalazine, at a dose not exceeding 3 g/day, provided that therapy was started at least 8 weeks before signing the ICF. Subjects with inflammatory bowel disease (IBD) may be treated with topical 5-aminosalicylic acid at therapeutic doses;

     * intra-articular and paraspinal glucocorticoids within 4 weeks prior to the Randomization Visit, intramuscular glucocorticoids within 2 weeks prior to the Randomization Visit;
     * use of alkylating agents at any time within 12 months prior to signing the ICF;
     * use of targeted synthetic disease-modifying antirheumatic drugs (kinase inhibitors) at any time before signing the ICF.
5. Vaccination with any vaccines within 12 weeks prior to signing the ICF.
6. Documented presence of one or more of the following conditions within 8 weeks before signing the ICF and during the screening period: acute anterior uveitis, exacerbated IBD (attack of Crohn's disease or exacerbation (relapse, attack) of ulcerative colitis), exacerbated psoriasis.

   Clarification: for subjects with IBD: IBD therapy must be stable for 8 weeks prior to signing the ICF. For subjects with psoriasis: topical products may be used.
7. A current diagnosis or a history of a severe immunodeficiency of any origin.
8. A diagnosis of HIV infection, hepatitis B, hepatitis C, syphilis.
9. The following laboratory test results at screening:

   * Transaminase (ALT and/or AST) activity >1.5 ULN;
   * ALP activity >1.5 ULN;
   * WBC count <3.0 cells×109/L;
   * Neutrophil count <1.5 cells× 109/L;
   * Lymphocyte count <0.8 cell×109/L;
   * Platelet count <100 cells×109/L;
   * Hemoglobin level <100 g/L;
   * Serum creatinine level >ULN.
10. A history of hypothyroidism/hyperthyroidism/autoimmune thyroiditis and/or abnormal TSH level at screening.
11. Active or latent tuberculosis, including a history thereof .
12. Major surgery within 4 weeks prior to signing the ICF or major surgery planned for the period of participation in the study.
13. Documented diagnosis of infectious mononucleosis within 8 weeks prior to signing the ICF and during the screening period, any active infection or recurrent infection within 4 weeks prior to signing the ICF and during the screening period, including fever ≥38 °C at the Randomization Visit; Clarification: if a subject presents with an acute infection during the screening, the screening can be extended if agreed with the Sponsor. In this case, the Sponsor's representative will decide whether the subject can be randomized. Subjects with body temperature ≥38 °C may be rescreened once 4 weeks after resolution of the condition.
14. A history of coronavirus infection (positive PCR test for SARC-CoV2-RNA) less than 14 weeks before signing the ICF.

    Clarification: including according to the subject.
15. A documented diagnosis of any other chronic infection that, in the opinion of the investigator, can increase the risk of infectious complications.
16. Severe infectious diseases (requiring hospitalization, parenteral use of antibacterial, antimycotic or antiprotozoal drugs) within 8 weeks prior to signing the ICF and during the screening period.
17. Systemic antibacterial, antimycotic or antiprotozoal therapy within 8 weeks prior to signing the ICF and during the screening period.
18. Epileptic seizures, a history of seizures.
19. A history of or current (at the time of signing the ICF and during the screening period) significant uncontrolled neuropsychiatric disorders, severe depression and/or suicide attempts, a risk of suicide and/or any psychiatric illness that, in the opinion of the investigator, may pose an excessive risk to the subject or have an impact on the subject's ability to follow the protocol.
20. Known (including from historical data) alcohol or drug dependence, psychoactive substance or drug abuse, evidence of alcohol/drug dependence or current abuse that, in the investigator's opinion, is a contraindication to AS therapy or limits treatment adherence.
21. The following diseases:

    * at screening and/or in the past and at the Randomization Visit: non-axSpA inflammatory joint disease (including rheumatoid arthritis, gout, psoriatic arthritis, Lyme disease, etc.),
    * at screening and/or at the Randomization Visit: reactive arthritis,
    * at screening and/or in the past and at the Randomization Visit: systemic autoimmune diseases (including systemic lupus erythematosus, systemic scleroderma, inflammatory myopathy, mixed forms of inflammatory connective tissue diseases, overlap syndrome, etc.).

    Exception: subjects with psoriasis who have not previously received and do not currently need systemic therapy, as well as patients with IBD regarded as an extraskeletal manifestation of axSpA, may be included in the study if all other eligibility criteria are met.
22. Comorbidities (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), including disorders ongoing at the time of screening, which, in the opinion of the investigator, may affect the course of radiographic axSpA, the results of assessment of its symptoms, or create an unacceptable risk to the subject from study therapy.
23. Grade 3 or 4 obesity.
24. Known allergy or intolerance to any component of the test drug, premedication drugs used in this clinical study.
25. A history of angioedema.
26. Fibromyalgia, or other conditions associated with chronic pain .
27. Lymphoproliferative diseases or malignancies with a remission duration of less than 5 years, with the exception of cured basal cell carcinoma and cervical cancer in situ .
28. Pregnancy, pregnancy planning (including pregnancy of female sexual partners of male study subjects) less than 8 weeks after the last administration of the test drug/placebo, breastfeeding.
29. Contraindications to MRI.
30. Simultaneous participation in other clinical studies, as well as previous participation in other clinical studies less than 3 months before signing the ICF, prior participation in this study.

Exception: subjects who dropped out of this study at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieved ASAS40 | week 24
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more

SECONDARY OUTCOMES:
Proportion of subjects with the ASDAS-CRP <1.3 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score <1.3
Proportion of subjects with the ASDAS-CRP ≥1.3 - <2.1 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score ≥1.3 - <2.1
Proportion of subjects with the ASDAS-CRP ≥2.1 - ≤3.5 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score ≥2.1 - ≤3.5
Proportion of subjects with the ASDAS-CRP >3.5 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Proportion of subjects with the Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) score >3.5
Proportion of subjects who achieved ASDAS-CII (clinically important improvement) | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Clinically important improvement defined as a decrease from baseline in ASDAS ≥1.1
Proportion of subjects who achieved ASDAS-MI (Major improvement) | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Major improvement (MI) defined as a decrease from baseline in ASDAS ≥2.0
ASDAS-CRP change from baseline | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Proportion of patients who achieved clinical response defined as an improvement of BASDAI by at least 50% compared to baseline; | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in BASDAI | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Proportion of subjects who achieved ASAS40 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more
Proportion of subjects who achieved ASAS20 | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more
Proportion of subjects who achieved ASAS5/6 | weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Ratio of patients who developed a response in at least 5 of 6 criteria of ankylosing spondylitis assessment score (ASAS)
Proportion of subjects who achieved ASAS partial remission | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in BASMI | weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Change from baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) score
Change from baseline in BASFI | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) score
Change from baseline in the swollen joint count (44 joints) | weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in MASES | weeks 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Change from baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Change from baseline in overall back pain severity (BASDAI No. 2) | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in nocturnal back pain severity | weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  Change from baseline in nocturnal back pain score during measured by Visual Analog Scale for Pain
Change from baseline in the quality of life assessed using EQ-5D-3L questionnaire | weeks 12, 24, 48, 108, 156
Change from baseline in SF-36 Physical Functioning compared to baseline | weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in SF-36 Mental Health compared to baseline | weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
Change from baseline in ASAS HI compared to baseline | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156
  ASAS Health Index
Change from baseline in SPARCC | weeks 24, 48, 108, 156
  Change from baseline in Spondyloarthritis Research Consortium of Canada Enthesitis (SPARCC)
Change from baseline in mSASSS | weeks 48, 108, 156
  Change from baseline in Modified stoke ankylosing spondylitis spinal score (nSASSS)
Proportion of subjects with adverse events | weeks 36, 160
Proportion of subjects with serious adverse events | weeks 36, 160
Proportion of subjects with grade 3 or higher adverse events according to CTCAE 5.0 | weeks 36, 160
Proportion of subjects prematurely withdrawn from the study due to adverse events | weeks 36, 160
Proportion of subjects with adverse events of special interest | weeks 36, 160

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Clinical Rheumatology Hospital №25, Saint Petersburg
  - North-Western state Medical University named after I.I. Mechnikov, Saint Petersburg